CLINICAL TRIAL: NCT01066039
Title: A Prospective, Multi-center, Open-label, Single Arm Study to Assess the Effect of Bisoprolol on Glycemic Level in Type II DIAbetic patieNTs With Suboptimal Blood Pressure Control (GIANT Study)
Brief Title: Phase 4 Study to Assess the Effect of Bisoprolol on Glycemic Level in Type II Diabetic Subjects With Suboptimal Blood Pressure Control
Acronym: GIANT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 200006-509
Record Dates: First submitted 2010-02-08; First posted 2010-02-10 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-06

CONDITIONS: Hypertension; Diabetes Mellitus, Type II
Keywords: Bisoprolol; Hypertension; Diabetes mellitus, Type II; Blood pressure; Glycemic level
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — Bisoprolol

ARMS (1):
- Bisoprolol (Experimental)
  Interventions: Drug: Bisoprolol

INTERVENTIONS:
Drug: Bisoprolol — Bisoprolol tablet will be administered orally at dose of 5 milligram (mg) once daily for 24 weeks. If the blood pressure is not less than 130/80 millimeter of mercury (mmHg) during the first 8 weeks of treatment (up-titration), then the dose will be adjusted to 10 mg daily. In cases of hypotensive effect, symptomatic bradycardia or arrhythmia, the daily dose will be reduced to 2.5 mg.
  Other Names: Concor; Concor Plus; ConcorCor; Lodoz

SUMMARY:
This is a 24-week, prospective, multicenter, open-label, single-arm study to assess the effect of bisoprolol on glycemic level in Type 2 diabetes mellitus (T2DM) controlled subjects with hypertension. The hypothesis of study is that there is no change in glycemic level and lipid metabolism as determined by glycosylated hemoglobin (HbA1c) using bisoprolol in T2DM subjects with suboptimal blood pressure (BP) control.

DETAILED DESCRIPTION:
Diabetes mellitus and hypertension are two of the most common chronic conditions, and each predisposes to accelerated atherosclerosis, cardiovascular disease, and death. There has been a concern that beta-blocker might have adverse effects in subjects with diabetes on glucose metabolism, but some data shows that highly beta-1 selective agents such as bisoprolol are essentially free of metabolic disturbances involving blood sugar, insulin sensitivity and lipids.

This is a prospective, multicenter, single-arm, open-label study to assess the glycemic effect of bisoprolol in T2DM subjects with suboptimal BP control.

After pre-screening period, each enrolled subject with T2DM and suboptimal BP control will undergo laboratory test for efficacy and safety measurement. After that, subject will continue his/her usual dosage of antihypertensive medication and bisoprolol will be added.

Subjects will be instructed to continue their diet and level of physical activity and to attempt to maintain current body weight until completion of the study.

Bisoprolol will be titrated upward until a dosage that lowers BP to less than 130/80 millimeter of mercury (mmHg) during the first 2 months of treatment. The maximum dosage of bisoprolol will be 10 mg once daily. Following 6 month of added bisoprolol therapy, all efficacy and safety measurements will be repeated.

The duration of study will be up to 24 weeks for each subject.

Objectives

Primary objective:

* To assess the effect of bisoprolol on glycemic control measured by change from baseline in HbA1c in T2DM subjects with suboptimal BP control

Secondary objectives:

* To evaluate the effects of bisoprolol, as add-on therapy, on BP in T2DM subjects with suboptimal BP control
* To evaluate the effects of bisoprolol, as add-on therapy, on insulin sensitivity as determined by Homeostasis Model Assessment-Insulin Resistance (HOMA-IR)
* To evaluate the effects of bisoprolol, as add-on therapy, on lipid metabolism as determined by lipid profile in T2DM subjects with suboptimal BP control
* To evaluate the safety and tolerability of bisoprolol in T2DM subjects with suboptimal BP control
* To assess the effects of bisoprolol combination therapy on insulin and c-peptide in T2DM subjects with suboptimal BP control compared to baseline
* To assess the effects of bisoprolol combination therapy on microalbumin and albumin/creatinine ratio in T2DM subjects with suboptimal BP control compared to baseline

ELIGIBILITY:
Inclusion Criteria:

* Age of 20 years or older and less than 80 years
* Subjects with T2DM
* Subjects who have failed to achieve an appropriate BP level as a result of treatment with any antihypertensive drug other than beta blockers - that is, with BP inadequately controlled to greater than or equal to (>=) 130/80 mmHg. However, those who have used a beta blocker before 12 weeks can be enrolled
* Subjects who underwent stable anti-diabetic regimen during the 12 weeks prior to screening
* Signed written informed consent

Exclusion Criteria:

* Ongoing insulin therapy
* Change in two HbA1c levels measured at an interval of 4 weeks or longer for the previous 6 months is at least 1% (the last HbA1c is measured within 4 weeks)
* Secondary hypertension
* Subjects with renal impairment (creatinine greater than 150 micromol per liter or 1.7 milligram per deciliter)
* Cardiovascular disease (uncontrolled or symptomatic arrhythmia, unstable angina, sick sinus syndrome, second or third degree atrioventricular (AV) block, bradycardia [less than 50 beats per minute], congestive heart failure, myocardial infarction, cerebral infraction attached within 12 weeks)
* Subjects requiring BP control by at least 3 different antihypertensive drugs, or with either systolic blood pressure (SBP) >=180 mmHg or diastolic blood pressure (DBP) >=110 mmHg at baseline
* Subjects with type 1 diabetes mellitus (T1DM)
* Uncontrolled diabetes with HbA1c >9%
* BMI >40 kilogram per square meter (kg/m^2)
* Pulmonary disease (chronic obstructive pulmonary disease [COPD], bronchial asthma)
* Other patients considered by the investigator to be not eligible for participation in this study for a legal or mental reason
* Contraindications for beta-blocker
* Pregnant or lactating women
* Use of an investigational drug within 30 days of entry to the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2010-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Ltd.
Locations (1):
- Seoul St. Mary´s Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Bisoprolol: Bisoprolol tablet was administered orally at dose of 5 milligram (mg) once daily for 24 weeks. If the blood pressure was not less than 130/80 millimeter of mercury (mmHg) during the first 8 weeks of treatment (up-titration), then the dose was adjusted to 10 mg daily. In cases of hypotensive effect, symptomatic bradycardia or arrhythmia, the daily dose was reduced to 2.5 mg.
Period: Overall Study
Arm/Group | Bisoprolol
Started | 202
Treated | 200
Completed | 158
Not Completed | 44
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 17
Not completed — Protocol Violation | 2
Not completed — Inclusion/Exclusion Criteria Violation | 9
Not completed — Investigator's Request | 1
Not completed — Dropout due to Insulin Administration | 1
Not completed — Additional Antihypertensive Required | 4
Not completed — Volunteer Failed to Make the Next Visit | 2
Not completed — Failure to Control Blood Pressure | 1
Not completed — Drug/Dose Adjustment Required | 1

BASELINE CHARACTERISTICS:
Population: Analysis population included all the participants who were enrolled in this study.
Groups:
- Bisoprolol: Bisoprolol tablet was administered orally at dose of 5 mg once daily for 24 weeks. If the blood pressure was not less than 130/80 mmHg during the first 8 weeks of treatment (up-titration), then the dose was adjusted to 10 mg daily. In cases of hypotensive effect, symptomatic bradycardia or arrhythmia, the daily dose was reduced to 2.5 mg.
Arm/Group | Bisoprolol
Number analyzed (Participants) | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92
  Male | 110

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Month 6
Description: HbA1c represents the percentage of glycosylated hemoglobin. The change in HbA1c at Month 6 was calculated as HbA1c at Month 6 minus HbA1c at baseline.
Time Frame: Baseline, Month 6
Population: Full analysis set (FAS) included all participants who received at least one dose of investigational product and for whom the primary efficacy endpoint (HbA1c) was measured.
Measure: Mean (Standard Deviation); unit: Percent HbA1c
Arm/Group | Bisoprolol
Number analyzed (Participants) | 175
Percent HbA1c
  Baseline | 6.79 (0.66)
  Change at Month 6 | 0.26 (0.64)

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Month 3
Description: HbA1c represents the percentage of glycosylated hemoglobin. The change in HbA1c at Month 3 was calculated as HbA1c at Month 3 minus HbA1c at baseline.
Time Frame: Baseline, Month 3
Population: FAS included all participants who received at least one dose of investigational product and for whom the primary efficacy endpoint (HbA1c) was measured.
Measure: Mean (Standard Deviation); unit: Percent HbA1c
Arm/Group | Bisoprolol
Number analyzed (Participants) | 175
Percent HbA1c | 0.15 (0.51)

3. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP) and Mean Blood Pressure (BP) at Month 6
Description: The change in SBP, DBP, and mean BP at Month 6 were calculated as SBP, DBP, and mean BP at Month 6 minus SBP, DBP, and mean BP at baseline, respectively. Mean BP was calculated using the formula: (DBP plus [{SBP minus DBP} divided by 3]).
Time Frame: Baseline, Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol
Number analyzed (Participants) | 175
mmHg
  SBP: Baseline | 147.8 (11.5)
  SBP: Change at Month 6 | -13.4 (15.4)
  DBP: Baseline | 89.0 (7.3)
  DBP: Change at Month 6 | -9.1 (9.0)
  Mean BP: Baseline | 108.6 (6.9)
  Mean BP: Change at Month 6 | -10.5 (10.2)

4. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) at Months 3 and 6
Description: HOMA-IR is as an indicator of insulin resistance in participants with Type 2 diabetes mellitus and comorbid hypertension. HOMA-IR was derived from fasting plasma glucose (FPG) and fasting insulin (FI) using the formula: (FI [micro international units per milliliter {mcIU/mL}] * FPG [millimole per liter {mmol/L}]) divided by 22.5. The change in HOMA-IR at Months 3 and 6 was calculated as HOMA-IR at Months 3 and 6 minus HOMA-IR at baseline.
Time Frame: Baseline, Months 3 and 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcIU/mL * mmol/L
Arm/Group | Bisoprolol
Number analyzed (Participants) | 175
mcIU/mL * mmol/L
  Baseline | 2.3 (1.8)
  Change at Month 3 | 0.1 (1.8)
  Change at Month 6 | 0.4 (2.5)

5. Secondary Outcome: Change From Baseline in Insulin Level at Months 3 and 6
Description: The change in insulin level at Months 3 and 6 was calculated as insulin level at Months 3 and 6 minus insulin level at baseline.
Time Frame: Baseline, Months 3 and 6
Population: FAS included all participants who took the investigational product at least once and for whom the primary efficacy endpoint (HbA1c) was measured.
Measure: Mean (Standard Deviation); unit: mcIU/mL
Arm/Group | Bisoprolol
Number analyzed (Participants) | 175
mcIU/mL
  Baseline | 7.5 (4.8)
  Change at Month 3 | 0.2 (4.5)
  Change at Month 6 | 0.6 (6.0)

6. Secondary Outcome: Change From Baseline in C-Peptide Level at Months 3 and 6
Description: The change in C-peptide level at Months 3 and 6 was calculated as C-peptide level at Months 3 and 6 minus C-peptide level at baseline.
Time Frame: Baseline, Months 3 and 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Bisoprolol
Number analyzed (Participants) | 175
nanogram per milliliter (ng/mL)
  Baseline | 2.3 (0.9)
  Change at Month 3 | 0.1 (0.8)
  Change at Month 6 | 0.2 (1.0)

7. Secondary Outcome: Change From Baseline in Total Cholesterol, Low Density Lipoprotein (LDL) Cholesterol, High Density Lipoprotein (HDL) Cholesterol and Triglyceride Level at Month 6
Description: The change in total cholesterol, low density lipoprotein (LDL) cholesterol, high density lipoprotein (HDL) cholesterol, and triglyceride levels at Month 6 was calculated as total cholesterol, LDL cholesterol, HDL cholesterol, and triglyceride levels at Month 6 minus total cholesterol, LDL cholesterol, HDL cholesterol, and triglyceride levels at baseline, respectively.
Time Frame: Baseline, Month 6
Population: FAS included all participants who took the investigational product at least once and for whom the primary efficacy endpoint (HbA1c) was measured. Here, "N" (number of participants analyzed) signifies those participants who were evaluable for this outcome measure and "n" signifies those participants who were evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Bisoprolol
Number analyzed (Participants) | 174
milligram per deciliter (mg/dL)
  Total Cholesterol: Baseline (n = 174) | 168.6 (32.3)
  Total Cholesterol: Change at Month 6 (n = 173) | -0.8 (26.3)
  LDL: Baseline (n = 174) | 93.3 (26.3)
  LDL: Change at Month 6 (n = 173) | -1.6 (22.5)
  HDL: Baseline (n = 174) | 49.2 (11.7)
  HDL: Change at Month 6 (n = 173) | -3.4 (8.0)
  Triglyceride: Baseline (n = 174) | 155.0 (96.3)
  Triglyceride: Change at Month 6 (n = 173) | 13.5 (87.6)

8. Secondary Outcome: Change From Baseline in Albumin/Creatinine Ratio at Month 6
Description: The change in albumin/creatinine ratio at Month 6 was calculated as albumin/creatinine ratio at Month 6 minus albumin/creatinine ratio at baseline.
Time Frame: Baseline, Month 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Bisoprolol
Number analyzed (Participants) | 89
ratio
  Baseline (n = 89) | 127.7 (630.9)
  Change at Month 6 (n = 85) | 34.3 (186.6)

9. Secondary Outcome: Change From Baseline in Microalbumin Level at Month 6
Description: The change in microalbumin level at Month 6 was calculated as microalbumin level at Month 6 minus microalbumin level at baseline.
Time Frame: Baseline, Month 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Bisoprolol
Number analyzed (Participants) | 167
mg/dL
  Baseline (n = 167) | 56.6 (261.6)
  Change at Month 6 (n = 161) | -3.1 (204.4)

10. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) was defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. A Serious Adverse Event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect.
Time Frame: Baseline up to Month 6
Population: Safety population included all participants who received at least one dose of investigational product.
Measure: Number; unit: participants
Arm/Group | Bisoprolol
Number analyzed (Participants) | 200
participants
  AEs | 68
  SAEs | 7

ADVERSE EVENTS:
Time Frame: Baseline up to Month 6
Arm/Group | Bisoprolol
Serious Adverse Events (participants affected / at risk) | 7/200
Other Adverse Events (participants affected / at risk) | 61/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bisoprolol (N=200)
Fracture lower limb (Musculoskeletal and connective tissue disorders) | 1
Fracture rib (Musculoskeletal and connective tissue disorders) | 1
Fracture upper limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gallbladder carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bisoprolol (N=200)
Oedema (General disorders) | 1
Oedema periorbital (General disorders) | 1
Pain legs (General disorders) | 1
Sensation of warmth (General disorders) | 1
Weakness generalized (General disorders) | 3
ECG abnormal (Cardiac disorders) | 1
AV block first degree (Cardiac disorders) | 1
Bradyarrhythmia (Cardiac disorders) | 1
Palpitation (Cardiac disorders) | 1
Dizziness (Nervous system disorders) | 6
Dizziness postural (Nervous system disorders) | 1
Headache (Nervous system disorders) | 8
Numbness (Nervous system disorders) | 2
Vocal cord paralysis (Nervous system disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 2
Enteritis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastritis aggravated (Gastrointestinal disorders) | 1
Gastritis atrophic (Gastrointestinal disorders) | 1
Gastro-intestinal disorder nos (Gastrointestinal disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
Gingivitis (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Periodontitis (Gastrointestinal disorders) | 1
Reflux oesophagitis (Gastrointestinal disorders) | 2
Tooth ache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Biliary stones (Hepatobiliary disorders) | 1
Liver fatty (Hepatobiliary disorders) | 1
Liver function tests abnormal nos (Hepatobiliary disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperlipaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2
Polydipsia (Metabolism and nutrition disorders) | 1
Weight decrease (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Jaw pain (Musculoskeletal and connective tissue disorders) | 1
Ligament disorder (Musculoskeletal and connective tissue disorders) | 1
Pain neck/shoulder (Musculoskeletal and connective tissue disorders) | 1
Larynx neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Insomnia (Psychiatric disorders) | 1
Anaemia (Investigations) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Common cold (Infections and infestations) | 3
Coryza (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1
Coughing (Respiratory, thoracic and mediastinal disorders) | 4
Dry cough (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sputum disorder (Respiratory, thoracic and mediastinal disorders) | 1
Throat pain (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Pruritus aggravated (Skin and subcutaneous tissue disorders) | 1
Skin injury (Skin and subcutaneous tissue disorders) | 1
Albuminuria (Renal and urinary disorders) | 1
Polyuria (Renal and urinary disorders) | 1
Renal cyst (Renal and urinary disorders) | 2
Peripheral coldness (Vascular disorders) | 1
Allergic conjunctivitis aggravated (Eye disorders) | 1
Cataract aggravated (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Eye abnormality (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No